CLINICAL TRIAL: NCT06840886
Title: An Open-label, Phase 1a/1b, Dose Escalation and Dose Expansion Study Investigating the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of PHST001 in Adult Patients With Advanced Relapsed and/or Refractory Solid Tumors
Brief Title: A Study of PHST001 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pheast Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PHST001-101
Record Dates: First submitted 2025-02-10; First posted 2025-02-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Dose levels are 0.1 mg/kg, 0.3 mg/kg, 1.0 mg/kg, 2.0 mg/kg, 4.0 mg/kg, 6.0 mg/kg, 9.0 mg/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Seven dose levels will be tested in dose escalation.
  Interventions: Drug: PHST001

INTERVENTIONS:
Drug: PHST001 — * PHST001 will be administered as IV infusions in a 3-week (Q3W) dosing interval. The dosing day will be on Day 1, 21 days cycle.
  * Other Names:
  * Dose Level 1
  * Dose Level 2
  * Dose Level 3
  * Dose Level 4
  * Dose Level 5
  * Dose Level 6
  * Dose Level 7
  Drug: PHST001
  * PHST001 will be administered as IV infusions in a 3-week (Q3W) dosing interval. The dosing day will be on Day 1, 21 days cycle.
  This study is an open label, Phase 1 dose escalation trial with three expansion cohorts. The study consists of two parts:
  * Part A: Dose escalation in patients with advanced solid tumors. Approximately 40-80 in total will be in enrolled in part A, covering 7 dose level.
  * Part B: Expansion cohorts will be added as an amendment as further preclinical data and clinical data from Part A become available.

SUMMARY:
PHST001-101 is a multicenter, open-label, Phase 1 study of PHST001 in patients with advanced solid tumors. The study design includes a Dose Escalation Phase and a Dose Expansion Phase, and will enroll patients with advanced relapsed and/or refractory solid tumors. The study's primary object is to evaluate the safety and tolerability of PHST001 and determine the RP2D (Recommended Phase 2 dose) of PHST001.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumor which has relapsed from or been refractory to all locally available standard therapies.
* Adequate hepatic function:
* AST and ALT ≤ 2.5 × times ULN (≤ 5 × ULN if liver metastases)
* Total bilirubin ≤ 1.5 × ULN (<3 ×ULN for patients with elevations due to Gilbert syndrome)
* Lipase and amylase ≤ 2×ULN
* Adequate renal function: calculated creatinine clearance of ≥ 30 mL/min calculated per institutional standard
* Adequate bone marrow function without packed RBC transfusion within the prior 2 weeks. Patients can be on a stable dose of erythropoietin (approximately ≥ 3 months). Criteria must be met without platelet transfusion within 7 days of screening blood draw:
* Absolute neutrophil count (ANC) ≥1,500/µL
* Platelet count ≥100,000/µL
* Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La

Key Exclusion Criteria:

* History of a previous additional malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 5 years. Patients with basal cell carcinoma of the skin, Stage I melanoma, melanoma in situ, squamous cell carcinoma of the skin, early-stage prostate cancer, or carcinoma in situ, excluding carcinoma in situ of the bladder, who have undergone potentially curative therapy are not excluded and can be enrolled regardless of disease-free period following completion of potentially curative therapy. Patients with early-stage breast cancer who have undergone curative intent treatment and with no disease recurrence for 2 years after treatment are not excluded.
* Active known CNS metastases and/or carcinomatous meningitis. Patients with previously treated CNS metastases may participate provided they are radiologically stable (ie, without evidence of progression for at least 2 weeks by repeat imaging [note that the repeat imaging should be performed during study screening]), clinically stable, and without requirement of steroid treatment for at least 14 days prior to the first dose of study treatment.
* Received prior systemic anticancer therapy including investigational agents within 21 days or, if shorter, within 5 half-lives prior to the first dose of study treatment. Patients must have recovered from all AEs due to previous therapies to Grade ≤1 or baseline. Patients with Grade ≤2 neuropathy may be eligible. Patients with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.
* Prior autologous or allogeneic hematopoietic stem cell transplant or solid organ transplant.
* Received previous treatment with another agent targeting CD24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
AE | 90 days after the last dose of PHST001
  Evaluate the safety and tolerability of PHST001
DLT | 21 days after the first dose of PHST001
  Evaluate the safety and tolerability of PHST001

SECONDARY OUTCOMES:
RECIST v1.1 | From screening and during treatment up to 2 years
  Assessment of preliminary antitumor activity of PHST001
PK | From treatment until 90 days after last dose of PHST001
  Cmax of PHST001
PD | From treatment until end of treatment of up to 2 years of PHST001
  RO (receptor occupancy) on peripheral neutrophils

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Duke Cancer Institute, Durham, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas